CLINICAL TRIAL: NCT03781869
Title: A Randomized Controlled Multicenter Clinical Trial to Compare the Efficacy and Safety of Anlotinib as the Maintenance Therapy for Extensive-stage Small Cell Lung Cancer After Combined With Etoposide and Cisplatin Chemotherapy
Brief Title: Study of Anlotinib as the Maintenance Therapy for Extensive-stage Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Dong Wang, chief physician, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALT-SCLC-01
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Extensive-stage Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; Anlotinib; Maintenance therapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Etoposide; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib + Chemotherapy (Experimental): Patients receive etoposide 100mg/m2 from day 1 to day 3, cisplatin 75mg/m2 on day 1, and Anlotinib 12mg/d on day 1 to day 14 , repeated every 21 days, a total of 4-6 cycles, and then continue to take Anlotinib 12mg/d on day 1 to day 14, repeated every 21 days until progressive Disease(PD).
  Interventions: Drug: Anlotinib Hydrochloride; etoposide and cisplatin
- Chemotherapy (Placebo Comparator): Patients receive etoposide 100mg/m2 from day 1 to day 3, cisplatin 75mg/m2 on day 1, repeated every 21 days, a total of 4-6 cycles, and then follow up observation until PD.
  Interventions: Drug: etoposide and cisplatin

INTERVENTIONS:
Drug: Anlotinib Hydrochloride; etoposide and cisplatin — etoposide 100mg/m2 from day 1 to day 3, cisplatin 80mg/m2 on day 1 and Anlotinib Day 1 to day 14 followed by 7 days off treatment in a 21-day cycle, repeated every 21 days
  Arms: Anlotinib + Chemotherapy
Drug: etoposide and cisplatin — etoposide 100mg/m2 from day 1 to day 3, cisplatin 80mg/m2 on day 1, repeated every 21 days
  Arms: Chemotherapy

SUMMARY:
Anlotinib has been approved as a third-line treatment for advanced non-small-cell lung cancer. A phase II clinical studies of small cell lung cancer (ALTER-1210) also showed that, compared with placebo, Anlotinib could improve the patients survival and had less toxic side effects after 2-3 line therapy. The purpose of this multicenter, randomized, prospective study is to investigate the efficacy and safety of Anlotinib as the maintenance therapy for Extensive-stage small cell lung cancer after combined with etoposide and cisplatin chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of small cell lung caner
* Advanced small cell lung cancer who had no prior cisplatin-based chemotherapy or radiotherapy,at least one measurable lesion (by RECIST1.1)
* Males or females between 18 Years to 75 Years.
* Performance status of 0～2 on the ECOG criteria.
* Main organs function is normal
* Expected survival is above three months.
* with asymptomatic brain metastases.
* At least one measurable lung tumor lesion (according to RECIST criteria, the application of conventional technology, diameter length of the lesion >= 20mm or spiral CT >=10mm).
* Adequate hematologic (Leukocyte count >= 4.0×109/L, neutrophil count>=2.0×109/L, hemoglobin>=95g/L, platelets>=100×109/L), hepatic function (aspartate transaminase (AST) & alanine transaminase(ALT)

  =<upper normal limit(UNL) x1.5, bilirubin level =< UNL x 1.5).
* Patient can take oral medicine.
* Patients have the ability to understand and voluntarily sign the informed consent, and allow adequate follow-up.

Exclusion Criteria:

* History of cardiovascular disease: congestive heart failure (CHF) > New York Heart Association (NYHA) II, active coronary artery disease(patients with myocardial infarction six months ago can be recruited), arrhythmias need to be treated (allow taking beta blockers or digoxin).
* Serious clinical infection (> NCI-CTCAE version 4.0 ,infection standard II).
* Patients with epilepsy who need to take medicine (such as steroids or anti epilepsy agents).
* The patients had accepted allogeneic organ transplantation.
* Bleeding tendency or coagulation disorders.
* patients who need renal dialysis.
* suffered from other tumor within 5 years( Except: cervical carcinoma in situ, cured basal cell carcinoma, cured bladder epithelial tumor).
* uncontrolled hypertension (systolic pressure>150 mmHg , or diastolic pressure> 90 mmHg).
* thrombosis or embolism(cerebrovascular accidents including transient ischemic attack within the last 6 months).
* pulmonary hemorrhage >CTCAE grade 2 within 4 weeks before first use of drugs.
* Other organ hemorrhage >CTCAE grade 3 within 4 weeks before first use of drugs.
* severe uncured wounds, ulcers or fracture.
* uncured dehydration.
* Drugs abuse and medical, psychological or social conditions may interfere with the patient's participation in research or the results of the evaluation effect.
* Patients are allergic to drugs used in research.
* Factors influencing the safety and compliance of patients.
* Inability to comply with protocol or study procedures.
* Pregnant or breast-feeding.
* The researcher believe that the Patient is not suitable to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From randomization，each 42 days up to PD or death(up to 24 months
  The first day of treatment to the date that disease progression is reported

SECONDARY OUTCOMES:
Overall survival | From randomization until death (up to 5 years)
  The first day of treatment to death or last survival confirm date
Objective Response Rate | each 42 days up to intolerance the toxicity or PD (up to 24 months)
Treatment-related adverse events | the first date of treatment to 30 days after the last dose of study drug,assessed up to 24 months
  Treatment-related adverse events are assessed by common terminology criteria for adverse events(CTCAE) V4.0.
Performance Status | the first date of treatment to 30 days after the last dose of study drug, assessed up to 24 months
  Performance Status of patients will be assessed by Zubrod-Eastern cooperative oncology group(ECOG)-world health organization(WHO).
Disease Control Rate | each 42 days up to intolerance the toxicity or PD (up to 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Dong Wang, PH.D, Principal Investigator — Daping Hospital, Third Military Medical University, Chongqing,China